CLINICAL TRIAL: NCT01016119
Title: Efficacy of Folrex in the Superior Extremity Rehabilitation After Acute Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Jose Luis Giroud Benítez, MINSAP
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-0915-CU
Record Dates: First submitted 2009-09-28; First posted 2009-11-18 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2010-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): In this group we will use Placebo cream, in the early rehabilitations in the upper extremity
  Interventions: Drug: Placebo
- Folrex (Experimental): In this group we will use Folrex cream, in the early rehabilitations in the upper extremity
  Interventions: Drug: Folrex

INTERVENTIONS:
Drug: Folrex — Folrex cream, in the early rehabilitations in the upper extremity, before daily rehabilitation
  Arms: Folrex
Drug: Placebo — Placebo cream, in the early rehabilitations in the upper extremity, before daily rehabilitation
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate whether Folrex, could improve the motor recovery of the upper extremity after stroke in comparison with placebo during 4 weeks of treatment.

DETAILED DESCRIPTION:
Periodical measures of the motor recovery, of the upper extremity, by Fugl-Meyer score, it will be done at the beginning, at fifth day and at month. Each value will be compare to evaluate whether the groups of patient improve.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute stroke < 24 hours.
* Patients with impairment up to 4 on NIHSS scale.
* Family support.
* Informed consent.

Exclusion Criteria:

* Presence of another disease not well controlled.
* Patient with dementia.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Periodical measures of the motor recovery, of the upper extremity, by Fugl-Meyer score, it will be done at the beginning, at fifth day and at month (4 weeks). | 4 weeks

SECONDARY OUTCOMES:
Barthel index | 4 weeks
National Institutes of Health Stroke Scale (NIHSS) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Salvador Allende Hospital, Havana, La Habana, Cuba